CLINICAL TRIAL: NCT00003697
Title: A Phase I Trial of 5, 6 Dimethyl Xanthenone - 4 - Acetic Acid (DMXAA) in Solid Tumors
Brief Title: Dimethylxanthenone Acetic Acid in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Glasgow (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066804; CRC-PHASE-I/II-PH1/048; EU-98065
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2009-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — vadimezan

INTERVENTIONS:
Drug: vadimezan

SUMMARY:
RATIONALE: Dimethylxanthenone acetic acid may stop the growth of cancer cells by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of dimethylxanthenone acetic acid in treating patients with solid tumors that have not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of dimethylxanthenone acetic acid (DMXAA) in patients with solid tumors. II. Establish a maximum tolerated dose for this drug in these patients. III. Determine the pharmacokinetics of DMXAA in these patients. IV. Determine the effect of this regimen on coagulation parameters, TNF and other cytokine production, nitric oxide, and serotonin production in these patients. V. Assess the efficacy of this drug in this patient population. VI. Determine the effect of this drug on tumor vasculature by evaluating any changes apparent on MRI scans in these patients.

OUTLINE: This is a dose escalation, multicenter study. Patients receive dimethylxanthenone acetic acid (DMXAA) IV over 20 minutes once weekly for 6 weeks, followed by 2 weeks of rest. An additional course of therapy may be administered in the absence of unacceptable toxicity or disease progression. Cohorts of 3 patients receive escalated doses of DMXAA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: A minimum of 3 patients will be accrued to each dose level used to determine the maximum tolerated dose.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed solid tumor that is not amenable to any standard therapy or is refractory to conventional therapy Tumor mass larger than 3 cm accessible to MRI scan Documented progression within the past 2 months

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: WHO 0-2 Life expectancy: Greater than 3 months Hematopoietic: Hemoglobin at least 9 g/dL WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.2 mg/dL ALT less than 2 times upper limit of normal (ULN) Alkaline phosphatase less than 2 times ULN Renal: Creatinine less than 1.5 mg/dL Other: Fertile patients must use effective contraception No concurrent malignancy except cone biopsied carcinoma in situ of the cervix and adequately treated basal or squamous cell carcinoma of the skin No other serious medical condition No uncontrolled infection or serious infection within the past 28 days Must live within 1 hour of Mount Vernon Hospital, UK

PRIOR CONCURRENT THERAPY: At least 4 weeks since prior anticancer therapy (6 weeks for nitrosoureas and mitomycin) and recovered

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 1995-10; Study Completion 1998-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon J.S. Rustin, MD, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (1):
- Mount Vernon Hospital, Northwood, England, United Kingdom

REFERENCES:
- [Background] Jameson MB, Sharp DM, Sissingh JI, Hogg CR, Thompson PI, McKeage MJ, Jeffery M, Waller S, Acton G, Green C, Baguley BC. Transient retinal effects of 5,6-dimethylxanthenone-4-acetic acid (DMXAA, ASA404), an antitumor vascular-disrupting agent in phase I clinical trials. Invest Ophthalmol Vis Sci. 2009 Jun;50(6):2553-9. doi: 10.1167/iovs.08-2068. Epub 2009 Apr 22. PMID 19387077
- [Result] Rustin GJ, Galbraith S, Taylor N, et al.: Impact on tumour perfusion measured by dynamic magnetic resonance imaging (MRI) in the phase I trial of 5,6-dimethyl xanthenone-4-acetic acid (DMXAA). [Abstract] Ann Oncol 9 (suppl 2): A-483, 126, 1998.
- [Result] Jameson M, Thompson P, Baguley B, et al.: Comparative pharmacokinetics and plasma protein binding of the novel anti-cancer agent 5,6-dimethylxanthenone-4-acetic acid in humans and mice. [Abstract] Proceedings of the American Society of Clinical Oncology A-746, 1997.